CLINICAL TRIAL: NCT01791036
Title: Postoperative Analgesia Produced by Adductor Canal (Distal Femoral Artery Compartment) Block Is Not Inferior to Femoral Nerve Block In Outpatient Arthroscopic Anterior Cruciate Ligament Repair
Brief Title: Adductor Canal Block In Anterior Cruciate Ligament (ACL) Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-5231-B
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Neuromuscular Block
Keywords: Adductor canal block; Femoral Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor Canal Block Group (Experimental): Adductor Canal Block
  Interventions: Procedure: Adductor Canal Block
- Femoral Nerve Block Group (Active Comparator): Femoral Nerve Block
  Interventions: Procedure: Femoral Nerve Block

INTERVENTIONS:
Procedure: Adductor Canal Block — Examination of the adductor canal using ultrasound will be performed using a high frequency linear probe. Following this the ultrasound probe will be positioned perpendicular to the skin in the medial upper-thigh region. The ultrasound probe will be moved either cephalad or caudad from its initial position in order to visualize the femoral artery immediately deep to the middle of the sartorius muscle. This point will then be selected as the appropriate level for needle insertion. Sham blocks using subcutaneous injection of normal saline will be used in both groups to maintain patient blinding.
  Arms: Adductor Canal Block Group
Procedure: Femoral Nerve Block — Examination of the femoral nerve using ultrasound will be performed using a high frequency linear probe. Following this the ultrasound probe will be positioned perpendicular to the skin at the level of the femoral crease. The femoral artery will be identified and the femoral nerve will then be located immediately lateral to the artery, deep to the fascia iliaca and superficial to the iliopsoas muscle. The needle will be positioned next to the femoral nerve. Following this 20 ml of 0.25% bupivacaine with epinephrine will be injected incrementally over a 1 to 2 minute period. Sham blocks using subcutaneous injection of normal saline will be used in both groups to maintain patient blinding.
  Arms: Femoral Nerve Block Group

SUMMARY:
Adductor canal block will provide adequate analgesia to patients undergoing arthroscopic ACL reconstruction surgery, yet result in less motor blockade than a femoral block.

DETAILED DESCRIPTION:
This study is designed to demonstrate that postoperative analgesia produced by the adductor canal block is not inferior to that produced by femoral nerve block in patients undergoing arthroscopic ACL reconstruction surgery. The study will also compare the degree of motor blockade of the adductor canal block to that of the femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists(ASA)classification I-III, Patients 18 to 50 years of age, BMI 18 - 40. Patients scheduled for anterior cruciate ligament reconstruction surgery under general anesthesia and nerve blocks.

Exclusion Criteria:

Refusal or inability to provide informed consent. Any contraindication to regional anesthesia including coagulopathy or bleeding diathesis, allergy to local anesthetics, infection, nerve injury or malignancy at the site of the block.

History of alcohol/drug dependence. History of long term opioid intake or chronic pain disorder. History of preexisting neuropathy in the operative leg History of significant psychiatric conditions that may affect patient assessment.

Inability to understand the informed consent and demands of the study. Allergy to any of the components of the multimodal analgesic regimen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  Postoperative cumulative opioid consumption during the first 24 hours. All doses of supplemental (PRN) oral and parenteral opioid analgesics required will be converted into equivalent doses of oral morphine
Motor Blockade | 30 minutes
  The degree of motor blockade 30 minutes following the block procedure
Pain Scores | 12,24 and 48 hours
  Visual Analog Pain scores at rest and with movement at admisssion and discharge from post-anesthesia care unit (PACU), AT DISCHARGE FROM same day surgery unit (SDC) and at 12, 24 and 48 hours

SECONDARY OUTCOMES:
Sensory blockade | 30 min
  The degree of sensory blockade 30 minutes following the block procedure
Spread of local anesthetic | 30 min
  Spread of local anesthetic from the injection site

OTHER OUTCOMES:
Block procedure time | min
  Block procedure time from probe placement on the skin to time of needle exit
Block success | 30 min
  1 or 0 on both sensory and motor block testing after 30 min for success

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — University of Toronto; Richard Brull, MD, Principal Investigator — UHN - Women's College Hospital and Toronto Western Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Williams BA, Kentor ML, Vogt MT, Irrgang JJ, Bottegal MT, West RV, Harner CD, Fu FH, Williams JP. Reduction of verbal pain scores after anterior cruciate ligament reconstruction with 2-day continuous femoral nerve block: a randomized clinical trial. Anesthesiology. 2006 Feb;104(2):315-27. doi: 10.1097/00000542-200602000-00018. PMID 16436852
- [Background] Dauri M, Fabbi E, Mariani P, Faria S, Carpenedo R, Sidiropoulou T, Coniglione F, Silvi MB, Sabato AF. Continuous femoral nerve block provides superior analgesia compared with continuous intra-articular and wound infusion after anterior cruciate ligament reconstruction. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):95-9. doi: 10.1097/AAP.0b013e31819baf98. PMID 19282706
- [Background] Sakura S, Hara K, Ota J, Tadenuma S. Ultrasound-guided peripheral nerve blocks for anterior cruciate ligament reconstruction: effect of obturator nerve block during and after surgery. J Anesth. 2010 Jun;24(3):411-7. doi: 10.1007/s00540-010-0916-3. Epub 2010 Mar 12. PMID 20225073